CLINICAL TRIAL: NCT03035240
Title: Finances First: A Health Intervention in Low Income Single Mother Households. A Prospective, Randomized, Controlled Trial to Assess the Effect of Financial Education on Health Outcomes in Single Mother Households.
Brief Title: Finances First: A Health Intervention in Low Income Single Mother Households
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1011656-1
Record Dates: First submitted 2017-01-26; First posted 2017-01-27 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2020-10

CONDITIONS: Financial Stress
MeSH Terms: conditions — Financial Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Financial Education Intervention (Experimental)
  Interventions: Behavioral: Financial Education
- No Financial Education Intervention (No Intervention)

INTERVENTIONS:
Behavioral: Financial Education — Participants randomized to financial education will undergo a year long financial education. This involves 9 weeks of weekly classes followed by one on one coaching for a year.
  Arms: Financial Education Intervention

SUMMARY:
The purpose of this prospective, randomized, controlled three-year study is to compare the effect of a year-long financial education program versus usual care on health outcomes in single mother low income households.

ELIGIBILITY:
Inclusion Criteria:

* Unmarried
* Currently employed
* Annual salary must be less than 200% of the Federal Poverty Guideline
* Supporting at least one child at home
* Able to read and speak either English or Spanish

Exclusion Criteria:

* Currently abusing alcohol or recreational drugs
* Currently living in a domestic violence situation
* Pregnant or planning to become pregnant in the next year

Ages: 19 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identified women - this would include those that identify as women
Enrollment: 345 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Changes in Quality of Life as measured by the WHO QOL BREF survey | Baseline and one year later
  Changes in Quality of Life as measured by the WHO QOL BREF survey
Weight loss | Baseline and one year later
  The proportion of overweight or obese women that achieve a 5% or more reduction in weight

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Packard, PharmD, Principal Investigator — Professor; Nicole White, PharmD, Principal Investigator — Associate Professor
Locations (1):
- Creighton University, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be shared with local Creighton Investigators listed on the study and the ICF. Individual participant data will not be shared outside of Creighton University.